CLINICAL TRIAL: NCT02161484
Title: A Prospective, Randomized, Blinded, Controlled Study Evaluating the Efficacy of Continuous Lumbar Plexus Block With and Without Parasacral Block in Patients Undergoing Total Hip Replacement
Brief Title: Continuous Lumbar Plexus Block With and Without Parasacral Block in Patients Undergoing Total Hip Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The computer is crushed and all data is lost (IT was not able to recover it. Last data was collected 6.17.14)
Sponsor: Rita Merman (Other)
Responsible Party: Sponsor-Investigator, Rita Merman, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO13030184
Record Dates: First submitted 2014-06-02; First posted 2014-06-11 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis of Hip; Regional Anesthesia; Other Acute Postoperative Pain; Total Hip Arthroplasty; Peripheral Nerve Block; Lumbar Plexus Nerve Block; Parasacaral (Sciatic) Nerve Block
Keywords: Peripheral Nerve Block; Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Lumbar Plexus Block with Parasacral Nerve Block (Experimental): Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm. In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.
  A single shot parasacral (sciatic) nerve block will then be place under the ultrasound guidance. Ropivacaine 0.2% 9 ml will be injected.
  Interventions: Procedure: Continuous Lumbar Plexus Block; Procedure: Parasacral Nerve Block; Drug: Ropivacine 0.2%; Drug: Bupivacaine 0.0625%
- Lumbar Plexus Nerve Block (Active Comparator): Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm. In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.
  No sham/placebo parasacral (sciatic) blocks will be performed in this group.
  Interventions: Procedure: Continuous Lumbar Plexus Block; Drug: Ropivacine 0.2%; Drug: Bupivacaine 0.0625%

INTERVENTIONS:
Procedure: Continuous Lumbar Plexus Block — Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm. In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.
Procedure: Parasacral Nerve Block — A single shot parasacral (sciatic) nerve block will then be place under the ultrasound guidance. Ropivacaine 0.2% 9 ml will be injected.
  Other Names: Sciatic Nerve Block
  Arms: Continuous Lumbar Plexus Block with Parasacral Nerve Block
Drug: Ropivacine 0.2% — Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm.
Drug: Bupivacaine 0.0625% — In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.

SUMMARY:
The purpose of this research study is to evaluate the analgesic efficacy of adding a single shot parasacral (sciatic) nerve block to a continuous lumbar plexus block in patients undergoing total hip replacement.

DETAILED DESCRIPTION:
This prospective study is intended to assess the efficacy of placing a parasacral (sciatic) nerve block in addition to a lumbar plexus block for postoperative analgesia following total hip arthroplasty. Although the placement of a lumbar plexus block alone has become accepted as the standard of care at UPMC for postoperative analgesia following total hip arthroplasty, the addition of a parasacral (sciatic) nerve block may provide the advantage of blocking the superior gluteal nerve and nerve to the quadratus femoris which both supply small articular sensory branches to the posterior hip capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated an Informed Consent Form.
2. Subject is classified as a ASA (American Society of Anesthesiologists) status I-III
3. Subject is age 18- 75 years old.
4. Subject is having primary total hip arthroplasty
5. No contraindication to peripheral nerve catheter ( local infection or hypocoagulable state)
6. Patient willing to receive spinal anesthesia as operative anesthesia
7. No known drug allergies to study medications
8. Patients not expected to receive therapeutic anticoagulation in the postoperative period.

Exclusion Criteria:

1. Subject inability to provide adequate informed consent.
2. Age younger than 18 years or older than 75 years
3. Any contraindication to the placement of lumbar plexus catheter, including local infection, hypocoagulable state.
4. ASA (American Society of Anesthesiologists) physical status of IV or greater
5. Any chronic painful conditions
6. Preoperative opioid use
7. Coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06-17 (Actual); Study Completion 2014-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Merman, MD, Principal Investigator — UPMC Presbyterian Shadyside; Jacques E. Chelly, MD, PhD, MBA, Study Chair — UPMC Presbyterian Shadyside
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Ben-Ari AY, Joshi R, Uskova A, Chelly JE. Ultrasound localization of the sacral plexus using a parasacral approach. Anesth Analg. 2009 Jun;108(6):1977-80. doi: 10.1213/ane.0b013e3181a04d8e. PMID 19448235
- [Background] Ho AM, Karmakar MK. Combined paravertebral lumbar plexus and parasacral sciatic nerve block for reduction of hip fracture in a patient with severe aortic stenosis. Can J Anaesth. 2002 Nov;49(9):946-50. doi: 10.1007/BF03016880. PMID 12419722
- [Background] Morris GF, Lang SA, Dust WN, Van der Wal M. The parasacral sciatic nerve block. Reg Anesth. 1997 May-Jun;22(3):223-8. doi: 10.1016/s1098-7339(06)80005-2. PMID 9168212
- [Background] Wiegel M, Gottschaldt U, Hennebach R, Hirschberg T, Reske A. Complications and adverse effects associated with continuous peripheral nerve blocks in orthopedic patients. Anesth Analg. 2007 Jun;104(6):1578-82, table of contents. doi: 10.1213/01.ane.0000261260.69083.f3. PMID 17513661
- [Background] Ilfeld BM, Mariano ER, Madison SJ, Loland VJ, Sandhu NS, Suresh PJ, Bishop ML, Kim TE, Donohue MC, Kulidjian AA, Ball ST. Continuous femoral versus posterior lumbar plexus nerve blocks for analgesia after hip arthroplasty: a randomized, controlled study. Anesth Analg. 2011 Oct;113(4):897-903. doi: 10.1213/ANE.0b013e318212495b. Epub 2011 Apr 5. PMID 21467563
- [Background] Marino J, Russo J, Kenny M, Herenstein R, Livote E, Chelly JE. Continuous lumbar plexus block for postoperative pain control after total hip arthroplasty. A randomized controlled trial. J Bone Joint Surg Am. 2009 Jan;91(1):29-37. doi: 10.2106/JBJS.H.00079. PMID 19122076

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Lumbar Plexus Block With Parasacral Nerve Block: Experimental: Continuous Lumbar Plexus Block with Parasacral Nerve Block
  Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm. In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.
  A single shot parasacral (sciatic) nerve block will then be place under the ultrasound guidance. Ropivacaine 0.2% 9 ml will be injected.
- Lumbar Plexus Nerve Block: Arm: Active Comparator: Lumbar Plexus Nerve Block
  Lumbar plexus nerve block placement and activation: After subcutaneous infiltration of local anesthetic, 20 mL of Ropivacaine 0.2% will be injected; the catheter will be introduced for 5 cm past the needle tip and secured with steri strips and tegaderm. In PACU, the catheter will be connected to a pump of 0.0625% bupivacaine at 5 - 10 mL per hour at the discretion of the Acute Interventional Perioperative Pain Service (AIPPS). Additional 5mL boluses of 0.0625% bupivacaine will be given on demand once per hour prn.
  No sham/placebo parasacral (sciatic) blocks will be performed in this group.
Period: Overall Study
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Started | 5 | 5
Completed | 1 | 2
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (2.86) | 58.6 (7.67) | 57.7 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Assessment
Description: Postoperative pain assessments using a 11-point numerical rating during physical therapy and at rest. This pain scale ranges from 0, being no pain at all, up to 10 being the worst pain ever experience.
Time Frame: 6 hours after the start of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 5 | 5
units on a scale
  Pain at Rest | 2.6 (2.19) | 3.6 (1.67)
  Pain with Movement | 3.5 (1.67) | 5 (1.87)

2. Primary Outcome: Numeric Rating Scale (NRS) Pain Assessment
Description: as for outcome 1
Time Frame: 24 hours after the start of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 4 | 5
units on a scale
  Pain at Rest | 4.25 (2.75) | 2.2 (1.92)
  Pain with Movement | 7.25 (2.5) | 4.4 (0.89)

3. Primary Outcome: Numeric Rating Scale (NRS) Pain Assessment
Description: as for outcome 1
Time Frame: 48 hours after the start of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 1 | 2
units on a scale
  Pain at Rest | 1 (0) | 2 (1.14)
  Pain with Movement | 8 (0) | 5 (1.41)

4. Secondary Outcome: Number of Rescue Boluses Administered by Nurse (IV Dilaudid) Post Operatively
Time Frame: 48 hours after the start of the surgery
Population: Results were not collected per source documentation. Since the IRB has expired, data pertaining to medications cannot be extracted from the medical record retrospectively.
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Amount of Oxycodone for the First 48 h Post Operatively
Description: Including number of dose and mg).
Time Frame: 48 hours after the start of the surgery
Population: as for outcome 4
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Dilaudid or Opiate Equivalent Consumed (mg) Over 48 Hours Post Operatively
Time Frame: 48 hours after the start of the surgery
Population: as for outcome 4
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Nerve Block Boluses (Bupivacaine) Administered by the Nurse Post Operatively
Time Frame: 48 hours after the start of the surgery
Population: as for outcome 4
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Total Amount of Local Anesthetic in 48 Hours Post Operatively
Description: Combined amount of Bupivacaine Boluses + Continuous infusion in (cc)
Time Frame: 48 hours after the start of the surgery
Population: as for outcome 4
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Incidence of Complications (e.g. Frequency of Foot-drop).
Description: Complications such as drug toxicity, arrhythmia, bradycardia, hematoma, "Foot Drop", allergic reaction will be recorded
Time Frame: 48 hours after the start of the surgery
Measure: Number; unit: Number of complications
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
Number analyzed (Participants) | 5 | 5
Number of complications | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment until 48 hours post-operatively or discharge from the hospital, whichever occurs first
Description: In addition to regular monitoring, questionnaires were given at 48 hours post-operatively to assess drug toxicity signs such as: numbness, ringing in ears, vision problems, motor weakness, metallic taste, etc.
Arm/Group | Continuous Lumbar Plexus Block With Parasacral Nerve Block | Lumbar Plexus Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes